CLINICAL TRIAL: NCT02126436
Title: Acupuncture for the Treatment of Phantom Limb Syndrome: A Randomised Controlled Trial (Feasibility Study)
Brief Title: Acupuncture for the Treatment of Phantom Limb Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London South Bank University (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLP001
Record Dates: First submitted 2014-04-09; First posted 2014-04-30 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Phantom Limb Syndrome
Keywords: phantom limb pain; phantom limb sensation; acupuncture; randomised controlled trial
MeSH Terms: conditions — Phantom Limb | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Active Comparator): Eight treatments of acupuncture will be given to participants twice weekly over four weeks. A combination of body and auricular acupuncture will be given and treatment will be pragmatic.
  In addition the group will receive usual care (including physiotherapy, occupational therapy, medical intervention and any other intervention as deemed appropriate by clinical staff).
  Interventions: Other: Acupuncture; Other: Usual care
- Usual care (Other): The group will receive usual care (including physiotherapy, occupational therapy, medical intervention and any other intervention as deemed appropriate by clinical staff).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Acupuncture — Participants will receive a course of traditional Chinese acupuncture. Acupuncture will be pragmatic but strict guidelines will be adhered to including:
  using a combination of body and auricular acupuncture, treating the opposite limb to amputation and possibly the residual limb, using auricular acupuncture points such as shen men, sympathetic, points corresponding to the lower limb, using body acupuncture points around the stump (depending on tissue health and the patient), mirroring local and distal points by needling them on the opposite limb, points on the lower back taking a segmental approach to dermatomal pain, including points such as LI4 + LR3, LR3, GV20, SP10, electro-acupuncture may be used, retaining the needles for 20-30 minutes, treating twice weekly for four weeks.
  Arms: Acupuncture
Other: Usual care — The group will receive usual care (including physiotherapy, occupational therapy, medical intervention and any other intervention as deemed appropriate by clinical staff).

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of acupuncture for the treatment of phantom limb syndrome in lower limb amputees and pilot an acupuncture protocol. The study will be a comparative effectiveness study comparing acupuncture and standard care versus standard care alone and will be a randomised controlled trial using a mixed methods approach. The study hypothesis is a course of acupuncture will reduce the symptoms of phantom limb syndrome in lower limb amputees.

The study will be based the Amputee Rehabilitation Unit, London. Twenty lower limb amputees with phantom limb syndrome will be randomly assigned to either receive usual care or usual care plus acupuncture. Acupuncture intervention will include 8 treatments over 4 weeks and treatment will involve using both body and auricular acupuncture points. Usual care will include physiotherapy, occupational therapy, pharmacological intervention and other interventions as deemed appropriate by clinical staff.

An eleven point numerical rating scale will be the primary outcome measure in this study. Secondary outcome measures will include the Short Form McGill Pain Questionnaire 2, EQ-5D-5L, Hospital Anxiety and Depression Scale, Perceived Stress Scale, Insomnia Severity Index, Participant Global Impression of Change and information will also be obtained on rescue medication. A cheek swab will also be taken to explore potential subgroups of responders in relation to the genetic polymorphism of the glucocorticoid receptor. Outcomes will be recorded weekly for the duration of the study and one and three months post completion of the study. In order to identify protocol acceptability and acceptability of outcome measures five participants will be interviewed post completion of the study. Data will also inform feasibility such as recruitment rate, completion rate and reasons for dropout.

Data from this study will guide the development of a full randomised controlled trial.

DETAILED DESCRIPTION:
The feasibility study will be a comparative effectiveness study. A randomised controlled trial (RCT) using a mixed methods approach will be employed to evaluate the effect of acupuncture on phantom limb syndrome. The RCT will be an open pragmatic effectiveness trial, of parallel and fixed size design with usual care control. It will be unstratified, with balanced randomization (1:1). It will be conducted at the Amputee Rehabilitation Unit (ARU) at Lambeth Community Care Centre, London, UK. Quantitative data will be collected using standardised, validated outcome measures. Qualitative data will be collected post completion of the study through one to one semi-structured interviews.

Twenty participants will be approached and recruited whilst they are inpatients at the ARU. Those felt to meet the inclusion criteria will be identified by the key contact in the rehabilitation team. Potential participants will then be approached by the researcher, provided with verbal and written information about the study and be advised to take up to seven days to consider if they wish to participate in the study or not. No consent will be obtained at the time of providing information about the study.

Participants who consent to being involved in the study will be screened for eligibility and if eligible will be randomly assigned into either, usual care plus acupuncture (group A) or usual care only (group B). Randomisation and allocation concealment will be used to ensure against selection bias. A computer generated random numbers table will be used in this study and randomisation will be unstratified and balanced (1:1). Allocation concealment will be implemented using sequentially numbered, opaque, sealed envelopes. Randomisation and allocation concealment will be generated by a researcher not directly involved in the study.

As the study is pragmatic all groups will receive usual care. Usual care will include both medical intervention, physiotherapy / rehabilitation and any other intervention used at the ARU. Group A will receive usual care and a standard course of acupuncture (as already agreed with an expert panel of acupuncture practitioners). Group B will receive standard care only. The acupuncture intervention in this study will be pragmatic but strict guidelines will be adhered to within this pragmatic approach. These guidelines have been developed though current literature and a Delphi study with acupuncture practitioners and consists of some specific acupuncture points and points selected for that patient according to Chinese diagnosis. Acupuncture guidelines include:

* Using a combination of body and auricular acupuncture
* Treating the opposite limb to amputation and possibly also the residual limb
* Using auricular acupuncture points such as shen men, sympathetic, points corresponding to the lower limb
* Using body acupuncture points around the stump (depending on the health of the tissue and the patient), mirroring local and distal points by needling them on the opposite limb, and points on the lower back taking a segmental approach to dermatomal pain
* Including points such as; LI4 + LR3, LR3, GV20, SP10 and individual specific points according to specific symptoms
* Electro-acupuncture may be used
* Retaining needles for 20-30 minutes
* Treating twice weekly for four weeks

At the commencement of the study group A and group B participant baseline demographic data will be collected by the researcher and in group A, a full Traditional Chinese Medicine Assessment will be completed by the acupuncture practitioner administering treatment. In both groups initial outcome measures will also be completed at this time and a cheek swab taken. For the duration of the study outcome measures will be collected once weekly from both groups by the researcher. Outcome measures will also be collected one and three months post completion of the study to assess long term effects of acupuncture intervention. At these two time points participants will be posted questionnaires to complete and return to the researcher.

In order to identify protocol acceptability and acceptability of which outcomes are meaningful to participants and would potentially demonstrate the impact of acupuncture in future trials, five participants will be consulted post completion of the study. This phase of the study will take a qualitative approach comprising of one off semi-structured interviews. This approach was taken to allow participants time to develop accounts of issues important to them with the aim of generating detailed data. If participants are still inpatients at the ARU at time of interview the interviews will take place there. If participants have been discharged the interview will take place in the participant's home or at their follow up outpatient appointment.

Data analysis will test for within-patient and between group differences in measurements taken at the beginning of the study, during the study, at the end and one month and three months post completion of the study. An intention to treat approach will be taken. In order to include missing data it will be imputed using last observation carried forward (LOCF).

Analysis of primary outcome measure (numerical pain rating scale): As the numerical rating scale produces ordinal data, median and range values will be evaluated. Raw change and percentage change will be calculated. A 95% confidence interval will be used in this study. Statistical analysis will be performed to verify rejection of the null hypothesis with a P value of 0.05 selected as indicative of statistical significance. As the data is ordinal and of small sample size non-parametric tests will be used in analysis. (Non parametric tests should be used on small sample sizes as under these conditions it is hard to see if data is normally distributed). The non-parametric Mann Whitney U test will be used for analysis between groups. Difference between baseline and last observation scores will be analysed using Wilcoxon signed-ranks test. All analysis will be undertaken using SPSS Version 21 software.

Analysis of secondary outcome measures: As all secondary outcomes produce ordinal data they will be treated as the numerical rating scale reporting median and range values and using the nonparametric tests as listed above. A P value of 0.05 will be considered indicative of statistical significance.

Baseline characteristics: Categorical data (such as gender and ethnicity) will be shown as n (%). As the study is small it is expected that data will not be normally distributed and therefore continuous data (such as age and duration of PLSd) will be shown as median and range values. Categorical baseline characteristics will be analysed using Fisher's exact test (as the data is categorical / nominal and unrelated). Continuous data will be analysed using the Mann-Whitney U test. As with the outcome measures a P value of 0.05 will be selected as indicative of statistical significance.

Feasibility Study Specific: Compliance with the protocol will be examined through number counts on drop outs / nonattendance completion rates of outcome measures and deviation from protocol.

Qualitative data analysis: Framework analysis will be used to analyse data from the semi-structured interviews. NVIVO 10 software will be used in data analysis. Data analysis will be transparent, comparative and reflexive. Analysis will focus on the latent content of the text. Transcripts will be read until the researcher is completely familiar with the data. Data will be coded, and an analytical framework will be developed. Data will then be indexed to the analytical framework, charted and mapped.

Reporting: Consolidated Standards of Reporting Trials (CONSORT) guidelines will be adhered to when reporting. The STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA) comprises of a checklist that expands the generic content of the CONSORT statement to include information on acupuncture intervention and will also be used in this study. Information will be recorded on style of acupuncture, reason for treatment provided, extent to which treatment was varied, number of needle insertions per subject per session, names of points used, depth of insertion, response sought, needle stimulation, needle retention time, needle type (diameter, length, manufacturer or material), number of treatment sessions, frequency and duration of treatment sessions, details of any other intervention administered (e.g. lifestyle advise), settings and context of treatment, practitioners background, precise description and rationale for control.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or above, full cognitive ability and able to communicate in English, able to provide informed consent and written informed consent obtained, current inpatients at the ARU (at time of enrolment), traumatic or medical amputation of a lower limb (greater than toes), currently experiencing phantom limb syndrome (with a verbal rating score of >4/10) in a lower limb.

Exclusion Criteria:

Less than 18 years of age, poorly controlled epilepsy, severe haemophilia or other bleeding / clotting disorders, pacemaker (if using electro-acupuncture), undergoing or recently undergone chemotherapy or bone marrow transplant, cognitive impairment and / or unable to give consent or communicate in English, medically unwell or severe other health complications (as advised by the medical consultant in charge of the participant), congenital limb absence, pregnancy, any skin changes or removal of lymph nodes on the body, ear or scalp that would preclude placement of acupuncture needles, needle phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale | Change from baseline at four weeks
  An eleven point scale will be used. The scale will present the numbers 0-10 with a description at 0 of 'no pain' and a description at 10 of 'pain as bad as you can imagine'. Participants will be asked to rate their average phantom pain over the last week

SECONDARY OUTCOMES:
Change in Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) | Change from baseline at four weeks
Change in EQ-5D-5L | Change from baseline at four weeks
Change in Hospital Anxiety and Depression Scale (HADS) | Change from baseline at four weeks
Change in The Insomnia Severity Index (ISI) | Change from baseline at four weeks
Patient Global Impression of Change (PGIC) | At four weeks
Change in Perceived Stress Scale (PSS) | Change from baseline at four weeks
Change in Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) | Change from baseline at one month
Change in Short Form McGill Pain Questionnaire 2 (SF-MPQ-2) | Change from baseline at three months
Change in EQ-5D-5L | Change from baseline at one month
Change in EQ-5D-5L | Change from baseline at three months
Change in Hospital Anxiety and Depression Scale (HADS) | Change from baseline at one month
Change in Hospital Anxiety and Depression Scale (HADS) | Change from baseline at three months
Change in The Insomnia Severity Index (ISI) | Change from baseline at one month
Change in The Insomnia Severity Index (ISI) | Change from baseline at three months
Change in Perceived Stress Scale (PSS) | Change from baseline at one month
Change in Perceived Stress Scale (PSS) | Change from baseline at three months
Change in Numerical Rating Scale | Change from baseline at one month
Change in Numerical Rating Scale | Change from baseline at three months

OTHER OUTCOMES:
Information will be obtained on adverse effects | At week one, two, three and four
  Adverse events will be captured through open ended prompts at each intervention point with participants
Cheek swab | Collect at baseline (before intervention)
  A cheek swab will be taken at the same time as when collecting demographic data to explore potential subgroups of responders in relation to the genetic polymorphism of the glucocorticoid receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Robinson, PhD, Principal Investigator — London South Bank University
Locations (1):
- GSTFT Amputee Rehabilitation Unit, Lambeth Community Care Centre, Monkton Street, London, United Kingdom

REFERENCES:
- [Background] Hu, X., Trevelyan, E., Yang, G., Lee, M. S., Lorenc, A., Liu, J. and Robinson, N. (2014a) The effectiveness of acupuncture or TENS for phantom limb syndromeII: A narrative review of case studies, European Journal of Integrative Medicine, (in press).
- [Background] Hu, X., Trevelyan, E., Yang, G., Lee, M. S., Lorenc, A., Liu, J. and Robinson, N. (2014b) The effectiveness of acupuncture/TENS for phantom limb syndrome. I: A systematic review of controlled clinical trials, European Journal of Integrative Medicine, (in press).
- [Derived] Trevelyan EG, Turner WA, Summerfield-Mann L, Robinson N. Acupuncture for the treatment of phantom limb syndrome in lower limb amputees: a randomised controlled feasibility study. Trials. 2016 Oct 25;17(1):519. doi: 10.1186/s13063-016-1639-z. PMID 27782861
- [Derived] Trevelyan EG, Turner WA, Robinson N. Acupuncture for the treatment of phantom limb pain in lower limb amputees: study protocol for a randomized controlled feasibility trial. Trials. 2015 Apr 12;16:158. doi: 10.1186/s13063-015-0668-3. PMID 25873101